CLINICAL TRIAL: NCT01715363
Title: Feasibility of an Immediate Preoperative Chemotherapy Before Resection of Colorectal Cancer and Research of Gene Expressions Changes Induced in the Tumor, Predictive of Chemotherapy Efficiency
Brief Title: Feasibility of an Immediate Preoperative Chemotherapy Before Resection fo Colorectal Cancer
Acronym: PRIMM
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-003446-41; 2010/1676 (Other: Institut Gustave Roussy)
Record Dates: First submitted 2012-10-24; First posted 2012-10-26 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Patients With Colorectal Cancer With Unresectable Synchronous Metastasis in Whom Resection of the Primitive Tumour is Indicated
MeSH Terms: interventions — Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FOLFOX + surgery + FOLFOX (Experimental): * Systemic chemotherapy (modified FOLFOX 4) 48 hours before surgery
  * resection of the colorectal tumor during surgery
  * Resumption of FOLFOX within the month after surgery (post operative administration of 4 course of treatment and assessment of the response)
  Interventions: Drug: Oxaliplatin; Drug: Folinic Acid; Drug: Fluorouracile

INTERVENTIONS:
Drug: Oxaliplatin
Drug: Folinic Acid
Drug: Fluorouracile

SUMMARY:
The purpose of this study is to analyze the clinical tolerance of immediate preoperative chemotherapy in terms of toxicity and perioperative morbidity and mortality

ELIGIBILITY:
Inclusion Criteria:

* colorectal metastatic adenocarcinoma (stage IV) with unresectables, measurables and visibles secondary lesions
* primitive tumor must be operate
* patient age between 18 and 70
* OMS status performance < 2
* life expectancy > 12 weeks
* hematologic function : PNN >/= 1.5x10^9/L, platelets >/= 100x10^9/L
* hepatic function : bilirubin </= 1.5xLSN, AST and ALT </= 3xLSN, alcalin phosphatasis </= 3xLSN
* plasmatimic creatin </= 1.25xLSN
* No previous chemotherapy or pelvic radiotherapy
* men and women in age of procreate agreeing to use a contraception until 4 months after the end of treatment for women and until 6 months for men

Exclusion Criteria:

* nonmetastatic forms
* Colorectal tumor which requires preoperative radiotherapy
* nonmeasurable metastasis based on RECIST criteria
* previous chemotherapy for colorectal cancer
* previous irradiation of the primitive tumour
* specific indication against the treatment studied
* Patient considered as inoperable for physiological or carcinologic reasons
* Pregnant or breast feeding women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Clinical tolerance of immediate preoperative chemotherapy | Assess up to 30 days after surgery
  Clinical tolerance of immediate preoperative chemotherapy assessment is based on the post-operative complication rate in terms of morbidity and mortality.
  All the post-operative complications arising within 30 days after surgery will be registered and classified using the Clavien Dindo classification

CONTACTS AND LOCATIONS:
Overall Officials: Diane GOERE, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Institut Gustave Roussy, Villejuif, Val de Marne, France